CLINICAL TRIAL: NCT06502015
Title: Biomarkers of Neurological Autoimmune Diseases
Brief Title: Biomarkers in Autoimmune Disease of Nervous System
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Daishi Tian, Prof., Tongji Hospital
Other Study IDs: TJ-IRB202406068
Record Dates: First submitted 2024-06-18; First posted 2024-07-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Autoimmune Diseases of the Nervous System; Neuromyelitis Optica Spectrum Disorder; Multiple Sclerosis; Guillain-Barre Syndrome; Acute Disseminated Encephalomyelitis; Autoimmune Encephalitis; Stiff-Person Syndrome; Myasthenia Gravis; Chronic Inflammatory Demyelinating Polyradiculoneuropathy; Idiopathic Inflammatory Myopathies; Autoimmune Diseases
Keywords: Biomarker; Autoimmune Diseases of the Nervous System; Immune cell
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Neuromyelitis Optica; Multiple Sclerosis; Guillain-Barre Syndrome; Encephalomyelitis, Acute Disseminated; Stiff-Person Syndrome; Myasthenia Gravis; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Myositis; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, feces, lymph nodes, bone marrow and brain tissue etc.al
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- autoimmune disease: clinical diagnosis with autoimmune disease of central nervous system
  Interventions: Diagnostic Test: biomaker levels
- health control: age- and sex-matched control individuals
  Interventions: Diagnostic Test: biomaker levels

INTERVENTIONS:
Diagnostic Test: biomaker levels — this study will discover and validate novel biomarkers (including blood, feces, bone marrow and lymph nodes etc al) of various neurological autoimmune diseases

SUMMARY:
Neurological autoimmune diseases are a group of disorders characterized by the abnormal immune response attacking the nervous system, including the brain, spinal cord and peripheral nerves. These diseases exhibit high heterogeneity, diverse clinical presentations, and are challenging to diagnose and manage due to a lack of effective treatments. In this study, the investigators will recruit eight kinds of autoimmune diseases of nervous system including Neuromyelitis Optica Spectrum Disorder (NMOSD), Myasthenia Gravis (MG), Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP), idiopathic inflammatory myopathy (IIM), and multiple sclerosis (MS), autoimmune encephalitis (AE), Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease (MOGAD). Through this study, the investigators aim to discover biomarkers with high sensitivity, specificity, and stability, which can support early diagnosis, disease monitoring, and personalized treatment for neurological autoimmune diseases, thereby improving the quality of life and prognosis for patients.

DETAILED DESCRIPTION:
Autoimmune diseases of the nervous system are a type of disease in which the human immune system mistakenly attacks its own nervous system, causing damage to the structure and function of the nervous system. Its main pathogenic mechanism is that autoimmune cells, autoantibodies and other immune molecules directly or indirectly attack the nervous system. Autoimmune diseases of the nervous system can affect the central nervous system, peripheral nervous system and neuromuscular junction, leading to pathological changes such as neuronal or axonal damage, demyelination, and destruction of neuromuscular junction. Autoimmune diseases of the nervous system are relatively rare, with a wide range of damage and complex and diverse clinical manifestations. They have the characteristics of complexity of immune diseases and high mortality and disability of nervous system diseases. At present, the understanding of the disease is limited, and some diseases are difficult to diagnose. Globally, it is a major cause of disability in young and middle-aged people and can cause huge social and economic burdens. However, due to the lack of a series of relatively reliable prognostic predictors, it is impossible to carry out personalized immunotherapy to achieve the best therapeutic effect, and serious adverse events may occur. Proteomics, metabolomics, intestinal microorganisms and intestinal high-throughput targeted metabolomics, exosomes, miRNA sequencing, single-cell transcriptome sequencing and other detection methods and lymphocyte subsets have been hot topics in the study of various diseases in recent years. It has been found that abnormalities in the expression and function of certain genes, proteins, metabolites, miRNAs, intestinal flora and lymphocyte subsets are closely related to the occurrence and development of many diseases and the functional disability of patients, and have a good suggestive effect on prognosis judgment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis with autoinflammatory diseases of the nervous system, including: Neuromyelitis Optica Spectrum Disorder (NMOSD), Myasthenia Gravis (MG), Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP), idiopathic inflammatory myopathy(IIM), multiple sclerosis (MS), autoimmune encephalitis (AE), Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease (MOGAD), ect al.
* sex and age-matched healthy individuals

Exclusion Criteria:

* Known history of primary immunodeficiency (innate or acquired).
* Patients with severe central nervous system, pulmonary, or other systemic infections.
* Patients with secondary central nervous system demyelinating lesions, such as those caused by vasculitis, systemic lupus erythematosus, and Sjögren's syndrome.
* Patients with vascular (including hemorrhagic and ischemic), hereditary metabolic, neoplastic, or toxic diseases.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with neurological autoimmune disease admission to Department of Neurology and Neurosurgery, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology from June 1, 2024 - May 31, 2034.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 10 years
  Death during the follow-up in every single reason

SECONDARY OUTCOMES:
Autoimmune disease of any kind | 10 years
  Brain or spinal MRI scans will be used to detect the presence of any autoimmune disease, including multiple sclerosis, neuromyelitis optica spectrum disorder, acute disseminated encephalomyelitis, autoimmune encephalitis, Guillain-Barré syndrome, and myasthenia gravis.

OTHER OUTCOMES:
Accumulated total active MRI lesions | 10 years
  the number of accumulate total active MRI lesions after CT103A infusion
Expanded Disability Status Scale (EDSS) score | 10 years
  EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS is a scale for assessing neurologic impairment in multiple sclerosis (MS). It consists of 7 FS (visual FS, brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, and cerebral FS) which are used to derive EDSS score ranging from 0 (normal neurological exam) to 10 (death from MS). A negative change from baseline indicates improvement. A participant was considered to have a worsening in overall EDSS score of at least 2 if baseline EDSS score was 0, or at least 1 point if baseline EDSS score is 1 to 5, or at least 0.5 point if baseline EDSS score is 5.5 or more.
Modified Rankin Scale | 10 years
  Modified Rankin Scale (mRS) is a profoundly valid and reliable measure of disability and is broadly utilized for assessing stroke outcomes and degree of disability. A favorable outcome was characterized as mRS ranging from zero up to two, while unfavorable outcome ranging for 3 up to 6.
Visual acuity | 10 years
  Corrected visual acuity is determine by Snellen E chart held at a distance of 5 meters. Higher score indicates better vision.
Quantitative Myasthenia Gravis Score (QMG) | 10 years
  Quantitative Myasthenia Gravis Score (QMG) range from 0 to 3. The normal person scored 0 and the higher score represent sever clinical symptom.
Myasthenia Gravis Activities if Daily Living (MG-ADL) Score | 10 years
  The MG-ADL is an eight-question survey of symptom severity, with each response graded from 0 (normal) to 3 (most severe). Two questions concern ocular, three oropharyngeal, one respiratory, and two extremity functions. Cumulative MG-ADL scores range from 0 to 24
Inflammatory Neuropathy Cause and Treatment (INCAT) Score | 10 years
  The INCAT score comprises two parts, the arm score and the leg score. Based on a patient's level of impairment in their arms and legs, each part is scored between 0 and 5 points, resulting in an INCAT total score between 0 and 10.
Medical Research Council (MRC) muscle function Score | 10 years
  The MRC score system for testing and grading of muscle function aims to provide a standardized and objective way to assess muscle function. It ranges from 0 to 5.
Manual Muscle Testing (MMT) Score | 10 years
  For MMT score, 16 muscle groups/ motions will be tested (not individual muscles). 14 of these are tested bilaterally. The score range from 0 to 10. A score of 10 is normal and a score of 0 is the worst.
36-item Short Form Generic Health Survey (SF-36) score | 10 years
  SF-36 will used to understand the health related quality-of -life of the subjects after CT103A infusion. The eight health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions will be searched. These outcomes will be grouped as physical component summary and mental component summary. The norm data is 0-100, the health related quality of life is increases as the scores are increased. The average score is 50.
EuroQol-five dimensions (EQ-SD) score | 10 years
  Health status is measured with the EuroQuality of Life Five Dimensions (EQ-5D) after CT103A infusion, which includes five dimensions and is used to evaluate the quality of life of sepsis survivors. They are mobility, self-care, usual activities, discomfort or pain and depression or anxiety. Levels are coded 1-5 and a total score is then generated. Results for the demographic measured will be displayed as a percentage value.
Visual analogue scale (VAS) pain score | 10 years
  usual visual analog scale (VAS) of pain is used to evaluate pain after CT103A infusion (line from 0: no pain to 10:worst pain)
Changes of concentration( pg/mL) of cytokines | 10 years
  such as ferritin, CRP, IL-6 and procalcitonin) will be analyzed
Profiling of immune cell subtypes | 10 years
  Changes in immune cells (including proportion of CD3+ T cells, CD3+CD4+ T cells and CD3+CD8+ T cells, ratio of CD4+ T/CD8+T) in blood, CSF and other immune organs will be analyzed through flow cytometry and single cell sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Dai-shi Tian, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McPherson RC, Anderton SM. Adaptive immune responses in CNS autoimmune disease: mechanisms and therapeutic opportunities. J Neuroimmune Pharmacol. 2013 Sep;8(4):774-90. doi: 10.1007/s11481-013-9453-9. Epub 2013 Apr 9. PMID 23568718
- [Result] Stenager E. A global perspective on the burden of multiple sclerosis. Lancet Neurol. 2019 Mar;18(3):227-228. doi: 10.1016/S1474-4422(18)30498-8. Epub 2019 Jan 21. No abstract available. PMID 30679041
- [Result] Solomon AJ, Arrambide G, Brownlee WJ, Flanagan EP, Amato MP, Amezcua L, Banwell BL, Barkhof F, Corboy JR, Correale J, Fujihara K, Graves J, Harnegie MP, Hemmer B, Lechner-Scott J, Marrie RA, Newsome SD, Rocca MA, Royal W 3rd, Waubant EL, Yamout B, Cohen JA. Differential diagnosis of suspected multiple sclerosis: an updated consensus approach. Lancet Neurol. 2023 Aug;22(8):750-768. doi: 10.1016/S1474-4422(23)00148-5. PMID 37479377